CLINICAL TRIAL: NCT00113854
Title: Effect of Mannitol as Adjunct Therapy on the Clinical Outcome of Childhood Cerebral Malaria in Mulago Hospital: A Randomised Clinical Trial
Brief Title: Mannitol as Adjunct Therapy for Childhood Cerebral Malaria
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD200211/246
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-06

CONDITIONS: Cerebral Malaria
Keywords: cerebral; malaria; children; mannitol; adjunct; therapy; Uganda
MeSH Terms: conditions — Malaria, Cerebral; Malaria | interventions — Mannitol

INTERVENTIONS:
Drug: Mannitol

SUMMARY:
Cerebral malaria is a life-threatening complication of Plasmodium falciparum infection in African children and nonimmune travellers despite availability of quinine, the current drug of choice. Several reports have suggested that raised intracranial pressure (ICP) is a major cause of death among children with cerebral malaria. Mannitol, an osmotic diuretic, effectively lowers ICP and is used to treat post traumatic raised ICP. There have been some case reports of reduction in mortality and morbidity in African children with cerebral malaria following administration of mannitol, but as these were not randomized controlled trials it is difficult to evaluate their significance. This study seeks to establish whether a single dose of intravenous mannitol given to children with cerebral malaria will significantly reduce the coma recovery time.

DETAILED DESCRIPTION:
Cerebral malaria is a life-threatening complication of Plasmodium falciparum infection accounting for significant morbidity and mortality in African children despite availability of quinine, the current drug of choice. The case fatality ranges from 5 to 40% with almost 10% of survivors experiencing neurological sequelae.

Several reports have suggested that raised intracranial pressure (ICP) may be a feature of cerebral malaria. There is evidence of brain swelling on computer tomography, magnetic resonance imaging and at necropsy. It has been postulated that raised intracranial pressure can cause death by transtentorial herniation or by compromising cerebral blood flow. In fact, most children who died of cerebral malaria in a Kenyan study, had clinical signs compatible with transtentorial herniation and all those who had severe ICP (maximum ICP > 40mmHg) either died or survived with neurological sequelae.

Mannitol, an osmotic diuretic, effectively lowers ICP and is used to treat post traumatic raised intracranial pressure. There have been some case reports of reduction in mortality and morbidity in African children with cerebral malaria following administration of mannitol, but as these were not randomized controlled trials it is difficult to evaluate their significance. Currently the WHO contends that there is insufficient evidence for using mannitol as adjunct therapy for cerebral malaria.

A recent Cochrane review found no randomized or quasi-randomized controlled trial to support or refute the use of mannitol as adjunct therapy for cerebral malaria.

Hypothesis: A single dose of intravenous mannitol (1g/kg) given to children with cerebral malaria will reduce mean coma recovery time from 22.5 to 13.1 hours.

We calculated a sample size of 78 patients in each group for 90% power and 95% confidence. In the calculation, we assumed that the children receiving intravenous mannitol would have a mean coma recovery time of 13.1 (SD 18.5) hours and those receiving placebo would have a mean coma recovery time of 22.5 (SD 18.5) hours (42.3% effect size), according to a recent study by Aceng, Byarugaba and Tumwine in the same hospital.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 5 years admitted to the Mulago hospital acute care unit during the study period with cerebral malaria: (seizures and unarousable coma lasting more than 30 minutes after seizures have stopped, with asexual forms of P. falciparum on the blood film, with no other cause of coma) and whose carers gave informed consent.

Exclusion Criteria:

* Children with evidence of having received any sedation within two hours prior to admission to the acute care unit.
* Also exclude children with clinical signs of pulmonary congestion, or heart failure, or renal disease, or shock

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156
Dates: Start 2004-10; Study Completion 2005-05

PRIMARY OUTCOMES:
Coma recovery time (that is time from beginning of antimalarial treatment until patient has fully regained consciousness).

SECONDARY OUTCOMES:
Time taken to sit un supported
Time to begin oral intake
Duration of hospitalisation
Mortality
Proportion of children recovering with neurological sequelae

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics and Child Health, Makerere Medical School, Kampala, Kampala, Uganda

REFERENCES:
- [Background] Aceng JR, Byarugaba JS, Tumwine JK. Rectal artemether versus intravenous quinine for the treatment of cerebral malaria in children in Uganda: randomised clinical trial. BMJ. 2005 Feb 12;330(7487):334. doi: 10.1136/bmj.330.7487.334. PMID 15705690
- [Background] Newton CR, Crawley J, Sowumni A, Waruiru C, Mwangi I, English M, Murphy S, Winstanley PA, Marsh K, Kirkham FJ. Intracranial hypertension in Africans with cerebral malaria. Arch Dis Child. 1997 Mar;76(3):219-26. doi: 10.1136/adc.76.3.219. PMID 9135262
- [Background] Newton CR, Kirkham FJ, Winstanley PA, Pasvol G, Peshu N, Warrell DA, Marsh K. Intracranial pressure in African children with cerebral malaria. Lancet. 1991 Mar 9;337(8741):573-6. doi: 10.1016/0140-6736(91)91638-b. PMID 1671941
- [Background] Okoromah CA, Afolabi BB. Mannitol and other osmotic diuretics as adjuncts for treating cerebral malaria. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD004615. doi: 10.1002/14651858.CD004615.pub2. PMID 15495121
- [Derived] Namutangula B, Ndeezi G, Byarugaba JS, Tumwine JK. Mannitol as adjunct therapy for childhood cerebral malaria in Uganda: a randomized clinical trial. Malar J. 2007 Oct 24;6:138. doi: 10.1186/1475-2875-6-138. PMID 17958887